CLINICAL TRIAL: NCT02839915
Title: Leucovorin for the Treatment of Language Impairment in Children With Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: Emory University (Other); Harvard University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Richard Frye, Principal Investigator and Sponsor, Southwest Autism Research & Resource Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAS-NIH; R01HD088528 (NIH)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Language Impairment
MeSH Terms: conditions — Autism Spectrum Disorder; Language Disorders | interventions — Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Folinic Acid (Experimental): Subjects randomized to receive Folinic Acid will take Liquid levo-leucovorin via oral route. The target dose is 1 mg/kg/day with a maximum of 25 mg/day, divided in two daily doses. A two- to four-week supply of 15 ml vials will be dispensed in line with the visit schedule. With the exception of children in the lowest weight group (≥ 15 - < 20 kg) from days 1-14, parents will administer the prescribed dose twice a day at the same time each day.
  Interventions: Drug: Folinic Acid
- Placebo Control (Placebo Comparator): Subjects randomized to receive placebo will take placebo twice a day (Exception: children in the lowest weight group ( ≥ 15 - < 20 kg) will start once a day for Days1-13). The pattern of dose escalation will be the same as the active compound. After 12 weeks, the blind will not be broken and subjects will be offered treatment for a 12-week open-label extension phase.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Folinic Acid — Liquid levo-leucovorin via oral route. L-leucovorin is the active isomer.
  Other Names: Liquid levo-leucovorin
  Arms: Folinic Acid
Other: Placebo — Inactive placebo comparator
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to determine the effectiveness of folinic acid in the treatment of language problems in children with autism spectrum disorder. Folinic acid, also known as leucovorin, is approved by the U.S. Food and Drug Administration (FDA) to decrease side effects during cancer chemotherapy. Folinic acid may be helpful in treating language problems in children with autism spectrum disorder, but this is not known. Therefore, folinic acid is an investigational new drug for this study. Investigators will enroll a total of 134 participants across all three centers, over a 5 year period and participation will last between 12 and 24 weeks.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a heterogeneous neurodevelopmental disorder often with life-long consequences that affects young children during critical developmental periods. The Centers for Disease Control estimates that ASD affects as many as 14.7 per 1000 children (1 in 68). Despite the dramatic rise in the detected prevalence of ASD over the past two decades, no effective medical treatment has been developed to address core ASD symptoms (social communication and repetitive behavior), the closely associated problem of language impairment, or the underlying pathophysiology of ASD. Currently, the only accepted treatment for core ASD symptoms is behavior therapy, which may entail intensive one-on-one treatment over several years.

The purpose of this study is to determine the effectiveness of folinic acid in the treatment of language problems in children with autism spectrum disorder. Folinic acid, also known as leucovorin, is approved by the U.S. Food and Drug Administration (FDA) to decrease side effects during cancer chemotherapy. Folinic acid may be helpful in treating language problems in children with autism spectrum disorder, but this is not known. Therefore, folinic acid is an investigational new drug for this study.

The primary aims of this study are to evaluate the efficacy and tolerability of high-dose folinic acid for improving the closely associated symptoms of language impairment in children with autism spectrum disorder (ASD). Improvement in delayed language may also benefit the core ASD problem of social communication. The study will also focus on identification of biomarkers in pre-specified subgroups of children with ASD that may moderate positive response to folinic acid. The study model is that high-dose folinic acid will improve language and set the stage for improved social communication in children with ASD and moderate language impairment. To test whether folinic acid is superior to placebo, 134 children (age 5 to 17 yrs 6 months, inclusive) with ASD and moderate language will be randomly assigned to folinic acid or placebo for 12 weeks under double-blind conditions. The study team will also test whether abnormalities in folate-dependent pathways, such as dysfunctional transport of folate across the blood-brain barrier, will moderate positive response to folinic acid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ≥ 5 years and < 17 years 5 months of age;
* Weight ≥ 15 kg;
* DSM-5 diagnosis of Autism Spectrum Disorder as established by clinical assessment, corroborated by the Social Communication Questionnaire and the Autism Diagnostic Observational Schedule.
* A score < 80 on the Core Language score of the Clinical Evaluation of Language Fundamentals -4 (CELF)- 4 or the Second Edition of the CELF-Preschool test (CELF-P).
* Current Clinical Global Impression Severity score ≥ 4 on ASD + communication delay.
* IQ at least 40 as measured by the Leiter-3 or mental age at least 18 months as measured on the Receptive Language Scale of the Mullen.
* Stable educational plan (one month) with no planned changes in the intensity of treatment for 12 weeks. (Otherwise eligible subjects with anticipated changes in their school program in the near term will be invited to return when the transition has been accomplished.
* Stable speech therapy program in the community (one month) with no planned changes for 12 weeks.
* English is spoken in the home and at least one parent is able to read, write and speak English.
* Stable medication (no changes in past 6 weeks and no planned changes for the next 6 months (duration of the study).

Exclusion Criteria:

* IQ below 40 as measured by the Leiter-3 or below a mental age of 18 months on the Receptive Language Scale of Mullen. (N.B. subjects who test below 18 months of age, but are otherwise eligible, may be enrolled following a case review by the Steering Committee - e.g., child's uncooperative behavior resulted in a likely underestimate of intellectual ability);
* Is within the scorable range of the CELF-4 or CELF-P as detailed in the Language Algorithm;
* Current DSM-IV diagnosis requiring alternative pharmacotherapy, e.g., Major Depression, Bipolar Disorder, a psychotic disorder (based on clinical assessment assisted by the Child and Adolescent Symptom Inventory);
* Presence of serious behavioral problems (tantrums, aggression, self-injury) for which another treatment is warranted.
* Significant medical condition by history or by physical examination or lab tests that would be incompatible with the study drug.
* Children taking anticonvulsant medication for seizures.
* Children taking Bactrim (trimethoprim + sulfamethoxazole) because Bactrim can interfere with folate metabolism. Children who discontinue use of Bactrim for 2 months may be re-evaluated for the study. Caregivers will be advised not to use any of these medications during the trial.
* Children taking valproic acid or derivatives or lamotrigine for any purpose will be excluded because these drugs can interfere with folate metabolism. Caregivers will be advised not to use any of these medications during the trial.
* Children on mineral or vitamin supplements that exceed the Recommended Daily Allowance set by the IOM.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Evaluation of Language Fundamentals 4 (CELF-4) Score. | Screening, Week 12
  The Scale title is the "Clinical Evaluation of Language Fundamentals 4" which is abbreviated as CELF-4 as indicated in the title above. Higher Scores indicate better performance. The Minimum Scaled Score is 40 and the Maximum Scaled Score is 160. The CELF-4 will be administered for participants between > 6.6 and < 12.5 years of age. The CELF-4 is comprised of 4 subtests intended to identify language problems and can be used to track progress over time. Administration of the CELF takes 30-45 minutes. The Core-CELF score is a composite that includes receptive and expressive language. Using the tables in the manual, raw scores from the four subtests are compared to normative data by age. The population mean = 100 + 15.
Change in Clinical Evaluation of Language Fundamentals Preschool (CELF-P) score | Screening, Week 12
  The Scale title is the "Clinical Evaluation of Language Fundamentals Preschool" which is abbreviated as CELF-P as indicated in the title above. Higher Scores indicate better performance. The Minimum Scaled Score is 40 and the Maximum Scaled Score is 160. The CELF-P will be administered for participants between > 5.0 and < 6.5 years of age to obtain an estimate of expressive and receptive language skills (based on population mean of 100 +15). Administration of the Core CELF-P takes 20-30 minutes. To make the CELF-P match the CELF-4, one additional subtest on CELF-P called the Concepts and Following Directions was added (this subtest is included in the Core of the CELF-4, but not included in the Core CELF-P).

SECONDARY OUTCOMES:
Change in Clinician Global Impression for Improvement (CGI-I) Score | Up to 12 Weeks
  The CGI-I is a 7-point measure of overall symptomatic change compared to baseline that will be used as a key secondary outcome measure. Scores range from 1 (Very Much Improved) through 4 (Unchanged) to 7 (Very Much Worse). The CGI-I will be rated by a clinician who is blind to treatment assignment, and will not engage in discussion of adverse events and medication dose. Ratings of "Much Improved" or "Very Much Improved" on the CGI-I will be used to define positive response. Subjects who drop out will be rated as non-responders.

OTHER OUTCOMES:
Change in the age appropriate version of the CELF compared to the pre-treatment level in the open-label extension phase | Pre-treatment, and 24weeks (or early termination)
  Change in the age appropriate version of the CELF compared to the pre-treatment level will be evaluated
Change in folate gene expression | Pre-treatment, 12 weeks(optional), and 24weeks (or early termination)
  Change in folate gene expression will be assessed by blood RNA test
Change in in methylation | Pre-treatment, 12 weeks (optional), and 24weeks (or early termination)
  Change in in methylation will be assessed by blood DNA test (or saliva test if the blood sample was insufficient)
Change in Aberrant Behavior Checklist (ABC) Score | Up to 12 Weeks
  The ABC is a 58-item consisting five subscales: hyperactivity, irritability, social withdrawal, stereotypic behavior and inappropriate speech in children with developmental disabilities. A higher score indicates more frequent aberrant behaviors.
Home Situations Questionnaire- Modified for ASD (HSQ-ASD) | Up to 12 Weeks
  The HSQ-ASD is a parent-rated scale of child noncompliance. The parent reports on the child's difficulties with compliance in 24 everyday situations. Questions answered affirmatively are then rated on a 1 to 9 Likert scale, with higher scores indicating more severe noncompliance. The scale yields a count of "yes" responses (0 to 27) and a severity score (total of 1 through 9 for all "yes" responses, for a range of 0 to 216
Children's Yale-Brown Obsessive-Compulsive Scales-ASD (CYBOCS-ASD) | Up to 12 Weeks
  The CYBOCS-ASD is a modified version of the CYBOCS developed for use in children with Obsessive-Compulsive Disorder. Each item is scored from 0 (least symptomatic) to 4 (most symptomatic), yielding a Total score from 0 to 20. It has established reliability and validity65 and is sensitive to change

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, PhD, Principal Investigator — Rossignol Medical Center
Locations (4):
- United States (4):
  - Southwestern Research and Resource Center, Phoenix, Arizona
  - Children's Healtcare of Atlanta, Atlanta, Georgia
  - Harvard University, Lexington, Massachusetts
  - State University of New York, Downstate, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: Yes
National Database for Autism Research
Time Frame: Biyearly NDAR is updated
Access Criteria: Registered for NDAR Access

REFERENCES:
- [Background] Frye RE, Rossignol DA, Scahill L, McDougle CJ, Huberman H, Quadros EV. Treatment of Folate Metabolism Abnormalities in Autism Spectrum Disorder. Semin Pediatr Neurol. 2020 Oct;35:100835. doi: 10.1016/j.spen.2020.100835. Epub 2020 Jun 25. PMID 32892962
- [Background] Frye RE, Slattery JC, Quadros EV. Folate metabolism abnormalities in autism: potential biomarkers. Biomark Med. 2017 Aug;11(8):687-699. doi: 10.2217/bmm-2017-0109. Epub 2017 Aug 3. PMID 28770615
- [Background] Frye RE, Slattery J, Delhey L, Furgerson B, Strickland T, Tippett M, Sailey A, Wynne R, Rose S, Melnyk S, Jill James S, Sequeira JM, Quadros EV. Folinic acid improves verbal communication in children with autism and language impairment: a randomized double-blind placebo-controlled trial. Mol Psychiatry. 2018 Feb;23(2):247-256. doi: 10.1038/mp.2016.168. Epub 2016 Oct 18. PMID 27752075
- [Background] Frye RE, Delhey L, Slattery J, Tippett M, Wynne R, Rose S, Kahler SG, Bennuri SC, Melnyk S, Sequeira JM, Quadros E. Blocking and Binding Folate Receptor Alpha Autoantibodies Identify Novel Autism Spectrum Disorder Subgroups. Front Neurosci. 2016 Mar 9;10:80. doi: 10.3389/fnins.2016.00080. eCollection 2016. PMID 27013943
- [Background] Frye RE, Sequeira JM, Quadros EV, James SJ, Rossignol DA. Cerebral folate receptor autoantibodies in autism spectrum disorder. Mol Psychiatry. 2013 Mar;18(3):369-81. doi: 10.1038/mp.2011.175. Epub 2012 Jan 10. PMID 22230883